CLINICAL TRIAL: NCT04669275
Title: The Effect Of Telephone Counselıng On Paın And Sleep Qualıty In Patıents Wıth Gastrıtıs Who Are Traıned In Gastrıtıs Management
Brief Title: Telephone Counseling in the Education of the Patient With Gastritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Nedret Tekin Kaya, Researcher, Eskisehir Osmangazi University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Eskisehir Osmangazi
Record Dates: First submitted 2020-11-29; First posted 2020-12-16 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Telenursing
Keywords: Telephone consultation; Gastritis; Pain; Quality of sleep
MeSH Terms: conditions — Gastritis; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telephone counseling (Experimental): People receiving telephone counselling.
  Interventions: Behavioral: Telephone Counselıng
- telephone counselin (Experimental): People receiving telephone counselling.
  Interventions: Behavioral: Telephone Counselıng

INTERVENTIONS:
Behavioral: Telephone Counselıng — Telephone counseling

SUMMARY:
It is planned to investigate the effect of telephone counseling on pain and sleep quality in patients with gastritis who have received gastritis management training. The individuals who constitute the target group in the planned study will be determined through the records of patients diagnosed with gastritis who applied to the Internal Medicine Polyclinic of Çankırı State Hospital. The target group of this study are individuals over the age of 18 diagnosed with gastritis. In the study, 18 years and older, who have Gastritis, have pain and sleep problems; The sample of the study is that patients with hearing loss, visual impairment, inability to understand / speak Turkish, who do not have a communication problem to prevent or prevent education or to participate in the study, who can communicate by phone, who are literate, and who voluntarily participate in the study.

DETAILED DESCRIPTION:
ABSTRACT It is planned to investigate the effect of telephone counseling on pain and sleep quality in patients with gastritis who have received gastritis management training. The individuals who constitute the target group in the planned study will be determined through the records of patients diagnosed with gastritis who applied to the Internal Medicine Polyclinic of Çankırı State Hospital. The target group of this study are individuals over the age of 18 diagnosed with gastritis. In the study, 18 years and older, who have Gastritis, have pain and sleep problems; The sample of the study is that patients with hearing loss, visual impairment, inability to understand / speak Turkish, who do not have a communication problem to prevent or prevent education or to participate in the study, who can communicate by phone, who are literate, and who voluntarily participate in the study. Research data will be collected with 7 forms prepared by the researcher.1.form is the elucidated form of consent, 2.form is the Introductory Information Form for determining the socio-demographic characteristics of the individuals who will participate in the research.3.form is the Richards Campbell Sleep Scale. 4. form is the Pain Assessment Scale. 5. Form is the Upper Gastrointestinal System Symptom Severity Scale. 6.form is the Tele Nursing Form for Gastritis Symptoms.7. form is the Telephone Call Evaluation Form.The planned study is an experimental study.The sample will be calculated by power analysis. The study will include an initiative group, a control group. Patients in both the initiative and the control group will be met and informed about the study by the researcher via face-to-face interview after their written and oral consent has been obtained. The first five forms will be applied to the control group and all 8 forms will be applied to the experimental group. The sampling individuals in the experimental group will receive gastritis management training and telephone counseling, while the individuals in the second group will form the control group. In the experimental group, the effect of a comprehensive gastritis management training program and 4 phone counseling and sms reminders one day a week on sleep quality and stomach pain will be evaluated. Phone calls 1. Week 3. Week 5. week and 7. it is weekly and will be performed biweekly.In the control group, no attempt will be made other than the rank given by the doctor. However, when the study is finished, a training booklet will be provided. An email was sent to the experts for the gastritis management training booklet prepared based on the relevant literature. DİSCERN Measurement Tool has also been sent as an e-mail to evaluate together with the booklet. The intervention group will be trained on topics such as reducing gastritis complaints, improving sleep quality, rational drug use, damages of smoking and alcohol, coping with stress, and factors triggering gastritis. Phone calls are expected to be between 12.00-18.00 and approximately 15 minutes.A business card will be printed by the researcher to enable patients to easily access the researcher. During the phone calls, they will be told that they can call on the topics they need between 08:00-20:00 in the evening.The results of the study will be analyzed in computer environment with SPSS program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* People with gastritis, pain and sleep problems;
* Without hearing loss,
* Without visual impairment,
* Can speak Turkish,
* Able to communicate by phone,
* Literate
* Patients who voluntarily participated in the study.

Exclusion Criteria:

* Being under 18,
* Without gastritis,
* With hearing disabilities,
* With visual disabilities,
* Can not understand and speak Turkish,
* Unable to communicate by phone,
* İlliterate,
* Patients who did not agree to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Change in the Visual Analog Skala Pain Scale, according to the initial measurement | At the beginning and at the 7th week
  The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically to digital. Two end definitions of the parameter to be evaluated are written on both ends of a 100 mm line and the patient is asked to indicate where his condition is appropriate by drawing a line or by placing a point or pointing on this line. For example, I have no pain at one end for pain, very severe pain is written on the other end, and the patient marks his current state on this line. The length of the distance from the place where there is no pain to the point marked by the patient indicates the patient's pain.
Change in the Richards - Campbell Sleep Scale, according to the initial measurement | At the beginning and at the 7th week
  There is a chart scored from 0 to 100 for each sleep statement. In this chart, "0" corresponds to the worst case and "100" to the best case for each statement.
Change in upper Gastrointestinal Symptom Severity Scale according to initial measurement | At the beginning and at the 7th week
  Contains questions about the severity of symptoms related to the gastrointestinal problem. For each symptom, the number is chosen that best represents how severe that symptom has been in the past two weeks. 0 = No symptoms, 1 = very mild, 2 = Mild, 3 = Moderate, 4 = Severe; 5 = Very severe

CONTACTS AND LOCATIONS:
Overall Officials: Nedret Tekin Kaya, Principal Investigator — Researcher
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, informed consent form
Supporting Information: Study Protocol, ICF
Time Frame: for 5 years
Access Criteria: You can access it by clicking the link. https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

REFERENCES:
- [Derived] Tekin Kaya N, Orsal O. "The Effect of Tele-Nursing on Pain and Sleep in Patients With Gastritis". Pain Manag Nurs. 2025 Dec;26(6):e515-e523. doi: 10.1016/j.pmn.2025.06.006. Epub 2025 Jul 8. PMID 40634176